CLINICAL TRIAL: NCT07187674
Title: Single Arm, Prospective, Small Sample, Exploratory Clinical Study on the Neoadjuvant Treatment of Early High-risk Triple Negative Breast Cancer With HRD Positive With Iparomlimab and Tuvonralimab(QL1706)Combined With Olaparib and Paclitaxel
Brief Title: The Neoadjuvant Treatment of Early High-risk Triple Negative Breast Cancer With HRD Positive With Iparomlimab and Tuvonralimab Combined With Olaparib and Paclitaxel
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Jinsong Wang, Chief physician, Harbin Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IITGC-1645-0513
Record Dates: First submitted 2025-09-10; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Triple Negative Breast Cancer (TNBC)
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — olaparib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Iparomlimab and tuvonralimab combined with olaparib and paclitaxel (Experimental)
  Interventions: Drug: Iparomlimab and tuvonralimab combined with olaparib and paclitaxel

INTERVENTIONS:
Drug: Iparomlimab and tuvonralimab combined with olaparib and paclitaxel — The main objective of this study is to evaluate the tpCR of early high-risk TNBC with HRD positive treated with Iparomlimab and tuvonralimab combined with olaparib and paclitaxel as neoadjuvant therapy

SUMMARY:
Breast cancer is one of the most common malignant tumors in women, accounting for the first cancer-related death cause in women. In recent years, the incidence has gradually increased, and the trend is younger. In 2022, the estimated number of new cases of female breast cancer worldwide is 2.389 million, and the estimated number of deaths is 666000. Triple negative breast cancer (TNBC) refers to breast cancer that is negative for estrogen receptor, progesterone receptor and human epidermal growth factor receptor 2, accounting for about 10% - 20% of malignant breast tumors. . At present, chemotherapy is still the main means of clinical treatment of TNBC, but the heterogeneity of TNBC in molecular level, pathology and clinical characteristics leads to different sensitivity of patients to different chemotherapeutic drugs, especially the sensitivity of most elderly patients to chemotherapeutic drugs is not high, and the prognosis is poor.

The development of immunotherapy in the field of breast cancer has witnessed the continuous deepening of medical understanding of cancer treatment. In the past, breast cancer was often regarded as a "cold tumor" insensitive to immunotherapy, but with the deepening of research, immunotherapy gradually occupied an important position in the treatment of breast cancer. The ongoing research hopes to identify patients who may benefit more from immunotherapy according to their respective tumor immune microenvironment.

Its mechanism of action mainly includes two aspects: one is to restore the normal recognition and attack ability of the immune system to tumor cells and break the immune escape mechanism of tumor cells; The second is to stimulate a lasting immune response, so that the immune system can continuously monitor and clear tumor cells.

Therefore, this study intends to evaluate the efficacy and safety of Iparomlimab and tuvonralimab combined with olaparib and paclitaxel in the neoadjuvant treatment of early high-risk TNBC with HRD positive.

It is planned to enroll 20 subjects. After enrollment, the subjects will receive six cycles of combination therapy with olaparib and docetaxel. Take 3 weeks as a treatment cycle until the treatment termination event specified in the protocol occurs, and the subject will continue to conduct postoperative efficacy and safety visits after the end of treatment.

After neoadjuvant treatment, according to the routine treatment process of breast cancer, the subject will receive breast cancer surgery; After surgical treatment, according to the residual breast lesions of the patient, the attending physician and the subject will agree on the subsequent treatment plan.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily join this study and sign an informed consent form;
2. Women aged ≥ 18 years and ≤ 70 years with early breast cancer:According to the definition of the latest ASCO/CAP guidelines, triple negative breast cancer patients with T1cN1-2 or T2-4N0-2 stage confirmed by histopathology;
3. Subjects with HRD positive tumor tissue evaluation;
4. According to RECIST 1.1, there must be at least one measurable lesion;
5. ECOG score: 0 to 1;
6. Tumor tissue specimens that can be used for biomarker detection;
7. The function of important organs meets the following requirements (no blood components or cell growth factor drugs are allowed to be used within 14 days before the first medication):

   Absolute neutrophil count ≥ 1.5 × 10^9/L; Platelets ≥ 100 × 10^9/L; Hemoglobin ≥ 90 g/L; Serum albumin ≥ 30 g/L; Thyroid stimulating hormone (TSH) ≤ 1 × ULN (if abnormal, FT3 and FT4 levels should be examined simultaneously. If FT3 and FT4 levels are normal, they can be included in the group); Serum total bilirubin ≤ 1.5 × ULN; ALT and AST ≤ 2.5 × ULN; AKP≤ 2.5×ULN； Serum creatinine ≤ 1.5 × ULN;
8. Female patients with non-surgical sterilization or childbearing age need to use a medically approved contraceptive measure (such as intrauterine device, contraceptive pill or condom) during the study treatment period and within 3 months after the end of the study treatment period; ; And must be non lactation; For male patients whose partners are women of childbearing age, effective methods of contraception should be used during the trial and within 3 months after the last administration of trial drugs.

Exclusion Criteria:

1. There is any active autoimmune disease or history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyperthyroidism; patients with vitiligo or asthma in childhood have been completely relieved and do not need any intervention after adulthood can be included; asthma requiring medical intervention with bronchodilators cannot be included);
2. Currently using immunosuppressants or systemic hormone therapy for immunosuppression (with a dosage of >10mg/day of prednisone or other equally effective hormones), and still continuing to use them within 2 weeks prior to enrollment;
3. Severe allergic reaction to other monoclonal antibodies;
4. Known history or evidence of interstitial lung disease or active non infectious pneumonia;
5. Having other malignant tumors in the past 5 years or at the same time (except for cured skin basal cell carcinoma and cervical carcinoma in situ);
6. Have hypertension and can not be well controlled after antihypertensive drug treatment; Had hypertension crisis or hypertensive encephalopathy in the past;
7. There are cardiac clinical symptoms or diseases that are not well controlled, such as: (1) heart failure above NYHA grade 2 (2) unstable angina pectoris (3) myocardial infarction within 1 year (4) clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention (5) qtc>450ms (male); Qtc>470ms (female);
8. The urine routine showed that the urine protein was ≥ + +, and the 24-hour urine protein volume was confirmed to be >1.0 g;
9. Patients with active infection, unexplained fever ≥ 38.5 ℃ within 7 days before medication, or white blood cell count >15 × 10^9/l at baseline;
10. Have congenital or acquired immune deficiency (such as HIV infected persons); Hepatitis B surface antigen (HBsAg) positive and hepatitis B virus deoxyribonucleic acid (HBV DNA) ≥ 2000 iu/ml, or hepatitis C virus antibody positive;
11. Less than 4 weeks before the study medication or may be vaccinated with live vaccines during the study period;
12. Bilateral breast cancer;
13. According to the judgment of the investigator, the patient has other factors that may affect the results of the study or cause the forced termination of the study, such as alcohol abuse, drug abuse, other serious diseases (including mental illness) requiring combined treatment, serious laboratory abnormalities, accompanied by family or social factors, which will affect the safety of the patient.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2028-06-15 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Total Pathological Complete Response (tpCR) | 5 months
  No invasive cancer cells in breast and axilla（ypT0/is N0）

SECONDARY OUTCOMES:
Breast Pathological Complete Respons(bpCR) | 5 months
  According to the evaluation method recommended by the international breast collaboration group：There is no residual invasive carcinoma in the primary breast lesion and regional lymph nodes, or only carcinoma in situ (such as ductal carcinoma in situ) remains. If there are solitary tumor cells or micrometastases in lymph nodes, it is still judged as non PCR。
Objective Response Rate(ORR) | 12 months
  Objective response rates assessed according to RECIST 1.1 criteria
3-year Disease Free Survival | 40 months
  The 3-year survival of Wu Bing evaluated according to RECIST 1.1 criteria
Ratio of Residual Cancer Burden (RCB) 0-1 | 5 months
  The RCB index is calculated by measuring indicators such as the size of the tumor bed, cell density, the proportion of in situ cancer, and lymph node metastasis
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 40 months

OTHER OUTCOMES:
Exploratory endpoint：PD-L1 expression level | 5 months
  Judge according to CPS table
Exploratory endpoint：TILs level | 5 months
  The method used was to perform hematoxylin eosin (He) staining on tissue sections, and further distinguish them by the typical characteristics of different lymphocytes or immunohistochemistry (IHC)
Exploratory endpoint：Ki-67 index | 40 months
  Taking the proliferation index of 14% as the critical point, the larger the value, the higher the malignant degree
Exploratory endpoint：Proportion of cd8+t cells | 5 months
  Immunohistochemical staining and flow cytometry